CLINICAL TRIAL: NCT05139615
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Hemodynamic Effects, Safety, Tolerability, and Pharmacokinetics of APD418 in Subjects With Heart Failure With Reduced Ejection Fraction
Brief Title: A Study to Assess the Hemodynamic Effects, Safety, Tolerability, and Pharmacokinetics of Intravenous APD418 in Adult Participants With Heart Failure With Reduced Ejection Fraction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD418-201; C5061001 (Other: Alias Study Number); 2020-006131-10 (EudraCT Number)
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Acute Heart Failure With Reduced Ejection Fraction
Keywords: Heart failure with reduced ejection fraction; HFrEF; APD418; Acute Heart Failure (AHF)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- APD418 (Part A: Dose Cohort 1-5) (Experimental)
  Interventions: Drug: APD418
- APD418 (Part B: Dose Group 1 and 2) (Experimental)
  Interventions: Drug: APD418
- Placebo (Part A: Cohort 1-5 and Part B) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APD418 — Participants will receive a single dose of APD418 as an intravenous (IV) infusion.
  Arms: APD418 (Part A: Dose Cohort 1-5)
Drug: APD418 — Participants will receive a single dose of APD418 as an IV infusion.
  Arms: APD418 (Part B: Dose Group 1 and 2)
Drug: Placebo — Participants will receive a single dose of APD418 matching placebo as an IV infusion.
  Arms: Placebo (Part A: Cohort 1-5 and Part B)

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, and effect on cardiac function of intravenous APD418 in adult participants with heart failure with reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
This study has an adaptive design, in which dose escalation in Part A will inform dose expansion in Part B. Part A is a single-ascending dose, placebo-controlled study planned to consist of 5 cohorts evaluating 5 doses of APD418. Part B is a parallel-treatment group study planned to evaluate 2 doses of APD418 and placebo. Participants in Part A cannot participate in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Advanced chronic Heart Failure with Reduced Ejection Fraction (HFrEF), defined as left ventricular ejection fraction (LVEF) less than or equal to (≤) 35% at Screening, including documented history of HFrEF (LVEF ≤ 35%) for at least 4 months prior to Screening
* New York Heart Association Class II-IV
* Cardiac index ≤ 2.5 liters per minute per square meter (L/min/m^2) and pulmonary capillary wedge pressure ≥ 15 millimeters of mercury (mm Hg) at Day 1
* Body mass index 18.0 to 37.0 kilograms per square meter (kg/m^2), inclusive, and body weight < 150 kg at Screening and Day 1

Exclusion Criteria:

* Hemodynamically unstable at Day 1 or in the opinion of the Investigator likely to progress to becoming hemodynamically unstable during the course of the study
* Treated with carvedilol or at a dose higher than a total of 25 milligrams per day any time within 72 hours of Day 1 through the end of the in-clinic observation Post-dose Period.
* Receiving any mechanical (respiratory or circulatory) or renal support therapy at Screening or Day 1
* Systolic Blood Pressure ≤ 90 millimeter of mercury (mm Hg) or ≥ 160 mm Hg, or Heart Rate < 50 beats per minute (bpm) or > 110 bpm, at Screening or Day 1
* Recently treated with inotropic, intravenous (IV) vasoactive or IV diuretic therapy, or expected to require such therapy with these drugs any time from Day 1 through the end of study conduct.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (5):
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - UnityPoint Health - Methodist Hospital, Peoria, Illinois
  - UTHealth, Houston, Texas
  - Health Science Center Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
- Germany (3):
  - Immanuel Hospital Bernau Brandenburg Heart Center, Bernau bei Berlin, Brandenburg
  - Kerckhoff-Klinik Forschungsgesellschaft GmbH, Bad Nauheim
  - Universitatsmedizin Greifwald, Greifswald
- Greece (3):
  - Konstantinopouleio General Hospital of Nea Ionia - Patision ''Agia Olga'', Nea Ionia, Athens
  - Interbalkan European Medical Center, Pylaia, Thessaloniki
  - General University Hospital of Larissa, Larissa
- Poland (3):
  - American Heart of Poland S.A., Gniezno
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza-Radeckiego, Wroclaw
- Serbia (7):
  - Clinical Hospital Centre Zemun, Belgrade
  - University Clinical Centre of Serbia, Belgrade
  - Institute for Cardiovascular Diseases Dedinje, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Institute for Cardiovascular Diseases of Vojvodina, Kamenitz
  - Clinical Center of Kragujevac, Kragujevac
  - Healthcare Center Uzice, Užice

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD418-201

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in two parts (Part A and B); however, study was terminated during Part A due to a business decision by Sponsor and Part B was not initiated and no participants were enrolled in Part B.
Groups:
- Cohort 1- 0.17 mg/kg/hr APD418: Participants were administered a single dose of 0.17 milligrams per kilogram per hour (mg/kg/hr) (total dose of 1 mg/kg) APD418 as an intravenous (IV) infusion over a duration of 6 hours on Day 1 (Dosing Period) followed by an 18 to 24-hour in-clinic observation period.
- Cohort 1- Placebo; Cohort 2- Placebo: Participants were administered a single dose of matching placebo as an IV infusion over a duration of 6 hours on Day 1 (Dosing Period) followed by an 18 to 24-hour in-clinic observation period.
- Cohort 2- 0.5 mg/kg/hr APD418: Participants were administered a single dose of 0.5 mg/kg/hr (total dose of 3 mg/kg) APD418 as an IV infusion over a duration of 6 hours on Day 1 (Dosing Period) followed by an 18 to 24-hour in-clinic observation period.
Period: Overall Study
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Started | 4 | 3 | 11 | 4
Completed | 4 | 3 | 11 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo | Total
Number analyzed (Participants) | 4 | 3 | 11 | 4 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 8 | 1 | 13
  >=65 years | 2 | 1 | 3 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 4 | 0 | 5
  Male | 3 | 3 | 7 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 11 | 4 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 11 | 4 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change in Cardiac Index (CI) Measured by Right Heart Catheterization (RHC) From Baseline to End of Intravenous (IV) Infusion at 6 Hours
Description: Cardiac index (CI) is a hemodynamic parameter that relates the cardiac output (CO) from left ventricle in one minute to body surface area (BSA), thus relating heart performance to the body size of the participant. It was measured by RHC.
Time Frame: Baseline (within 2 hours prior to start of study treatment administration) up to 6 Hours (end of IV infusion)
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Liter per minute per meter square
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Liter per minute per meter square | 0.33 (0.660) | 0.10 (0.100) | 0.25 (0.372) | 0.10 (0.245)

2. Secondary Outcome: Part A: Change in Stroke Volume (SV), Left Ventricular End-Systolic Volume (LVESV) and Left Ventricular End-Diastolic Volume (LVEDV) Measured by Echocardiogram (ECHO) From Baseline to End of IV Infusion at 6 Hours
Description: SV is the volume of blood pumped from the left ventricle per beat. LVESV is the volume of blood in the left ventricle at the end of contraction and at diastole. LVEDV is the amount of blood in the heart's left ventricle just before the heart contracts. All these parameters were measured by ECHO.
Time Frame: Baseline (within 2 hours prior to start of study treatment administration) up to 6 Hours (end of IV infusion)
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment. Here, 'Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 1 | 9 | 4
Milliliter
  Stroke Volume | 3.13 (10.623) | -0.80 (NA) — Standard Deviation could not be calculated as a single participant was analyzed. | 5.94 (10.183) | -3.15 (7.152)
  LVESV | -11.05 (22.837) | 4.10 (NA) — Standard Deviation could not be calculated as a single participant was analyzed. | 8.28 (25.689) | 8.92 (29.804)
  LVEDV | -7.92 (15.531) | 3.30 (NA) — Standard Deviation could not be calculated as a single participant was analyzed. | 14.20 (31.021) | 7.30 (38.006)

3. Secondary Outcome: Part A: Change in Stroke Volume Index (SVI) Measured by ECHO From Baseline to End of IV Infusion at 6 Hours
Description: SVI was calculated as stroke volume divided by BSA. This was measured by ECHO.
Time Frame: Baseline (within 2 hours prior to start of study treatment administration) up to 6 Hours (end of IV infusion)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliliter per meter square
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 1 | 9 | 4
Milliliter per meter square | 1.50 (5.518) | -0.30 (NA) — Standard Deviation could not be calculated as a single participant was analyzed. | 2.62 (4.615) | -2.00 (4.492)

4. Secondary Outcome: Part A: Change in Left Ventricular Ejection Fraction (LVEF) Measured by ECHO From Baseline to End of IV Infusion at 6 Hours
Description: LVEF is the central measure of left ventricular systolic function. LVEF is the fraction of chamber volume ejected in systole (stroke volume) in relation to the volume of the blood in the ventricle at the end of diastole (end-diastolic volume). This was measured by ECHO.
Time Frame: Baseline (within 2 hours prior to start of study treatment administration) up to 6 Hours (end of IV infusion)
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Percentage of end diastolic volume
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Percentage of end diastolic volume | 1.90 (6.009) | 0.47 (1.457) | 1.14 (3.204) | -1.68 (0.900)

5. Secondary Outcome: Part A: Change in Fractional Shortening (FS) Measured by ECHO From Baseline to End of IV Infusion at 6 Hours
Description: FS was calculated by measuring the percentage reduction in left ventricular diameter during systole. This was measured by ECHO.
Time Frame: Baseline (within 2 hours prior to start of study treatment administration) up to 6 Hours (end of IV infusion)
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Percentage | -2.60 (7.791) | 0.47 (5.710) | -1.55 (1.924) | -4.50 (7.444)

6. Secondary Outcome: Part A: Change in Left Ventricular End-Systolic and Left Ventricular End-Diastolic Diameter Measured by ECHO From Baseline to End of IV Infusion at 6 Hours
Description: Left ventricular end-systolic diameter and left ventricular end-diastolic diameter were measured using ECHO.
Time Frame: Baseline (within 2 hours prior to start of study treatment administration) up to 6 Hours (end of IV infusion)
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Centimeter (cm)
  Left ventricular end-systolic diameter | 0.10 (0.361) | -0.04 (0.384) | 0.22 (0.321) | 0.35 (0.544)
  Left ventricular end-diastolic diameter | -0.04 (0.087) | -0.02 (0.098) | 0.15 (0.363) | 0.16 (0.243)

7. Secondary Outcome: Part A: Change in Left Ventricular Global Longitudinal Strain (LVGLS) and Left Ventricular Global Circumferential Strain (LVGCS) Measured by ECHO From Baseline to End of IV Infusion at 6 Hours
Description: Left ventricular global strain is the average strain of the cardiac chamber wall, where LVGLS presents longitudinal shortening as a percentage (change in length as a proportion to baseline length). LVGCS measures the chamber deformation along the circumference of the cardiac wall in a tangential xy-direction and similarly presents the circumferential shortening as a percentage. Both the parameters were measured by ECHO.
Time Frame: Baseline (within 2 hours prior to start of study treatment administration) up to 6 Hours (end of IV infusion)
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment. Here, 'Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 1 | 1 | 5 | 4
Percentage
  LVGLS: number analyzed (Participants) | 1 | 1 | 4 | 4
  LVGLS | 0.30 (NA) — Standard Deviation could not be calculated as a single participant was analyzed. | -1.10 (NA) — Standard Deviation could not be calculated as a single participant was analyzed. | 1.10 (1.337) | -1.29 (0.987)
  LVGCS: number analyzed (Participants) | 1 | 0 | 5 | 2
  LVGCS | -6.70 (NA) — Standard Deviation could not be calculated as a single participant was analyzed. |  | 0.05 (2.105) | 0.00 (3.111)

8. Secondary Outcome: Part A: Change in CI Measured by RHC at 0.5, 1, 2, 3, 4 and 5 Hours During 6 Hour IV Infusion
Description: CI is a hemodynamic parameter that relates the CO from left ventricle in one minute to BSA, thus relating heart performance to the body size of the participant. It was measured by RHC.
Time Frame: Baseline (within 2 hours prior to start of study treatment administration), 0.5, 1, 2, 3, 4 and 5 hours of IV infusion
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Liter per minute per meter square
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Liter per minute per meter square
  0.5 hours | -0.05 (0.252) | 0.27 (0.379) | 0.10 (0.167) | -0.10 (0.183)
  1 hour | 0.35 (0.252) | 0.27 (0.379) | 0.06 (0.112) | 0.05 (0.208)
  2 hours | 0.45 (0.370) | 0.13 (0.058) | 0.11 (0.104) | -0.08 (0.126)
  3 hours | 0.68 (0.427) | 0.20 (0.265) | 0.20 (0.279) | 0.15 (0.129)
  4 hours | 0.25 (0.100) | 0.10 (0.100) | 0.09 (0.221) | 0.10 (0.346)
  5 hours | 0.23 (0.457) | 0.17 (0.153) | 0.11 (0.274) | 0.08 (0.096)

9. Secondary Outcome: Part A: Change in Cardiac Output (CO) Measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 Hours
Description: Change in CO measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 hours during the 6-hour IV infusion was reported in this outcome measure.
Time Frame: Baseline (within 2 hours prior to start of study treatment administration), 0.5, 1, 2, 3, 4, 5 and 6 hours of IV infusion
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Liter per minute
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Liter per minute
  0.5 hours | -0.15 (0.420) | 0.63 (0.777) | 0.20 (0.329) | -0.15 (0.300)
  1 hour | 0.68 (0.457) | 0.67 (0.907) | 0.15 (0.230) | 0.13 (0.340)
  2 hours | 0.90 (0.876) | 0.43 (0.231) | 0.21 (0.212) | -0.08 (0.189)
  3 hours | 1.28 (0.877) | 0.47 (0.643) | 0.41 (0.568) | 0.33 (0.299)
  4 hours | 0.43 (0.222) | 0.27 (0.231) | 0.18 (0.467) | 0.20 (0.560)
  5 hours | 0.43 (0.911) | 0.43 (0.379) | 0.25 (0.559) | 0.15 (0.191)
  6 hours | 0.75 (1.420) | 0.30 (0.346) | 0.53 (0.742) | 0.23 (0.499)

10. Secondary Outcome: Part A: Change in Pulmonary Capillary Wedge Pressure (PCWP), Right Atrial Pressure (RAP), Systolic Pulmonary Arterial Pressure/Diastolic Pulmonary Arterial Pressure (PAS/PAD) Measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 Hours
Description: PCWP estimated the left atrial pressure and was the pressure measured by wedging a pulmonary artery catheter with an inflated balloon into a small pulmonary arterial branch. PCWP was assessed by 2 successive measurements at least 10 minutes apart. RAP is the blood pressure in the right atrium of the heart. Change in PCWP, RAP, PAS/PAD at 0.5, 1, 2, 3, 4, 5 and 6 hours during the 6-hour IV infusion was reported in this outcome measure. All the parameters were measured by RHC.
Time Frame: as for outcome 9
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment. All participants reported under 'Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' (n) signifies number of participants evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Millimeters of mercury
  PCWP: 0.5 hours: number analyzed (Participants) | 4 | 3 | 9 | 3
  PCWP: 0.5 hours | 1.50 (2.887) | 0.67 (3.055) | -0.78 (3.456) | -2.67 (4.726)
  PCWP: 1 hour: number analyzed (Participants) | 4 | 3 | 9 | 3
  PCWP: 1 hour | -0.25 (8.808) | -2.33 (4.041) | -2.00 (2.828) | -2.67 (8.145)
  PCWP: 2 hours: number analyzed (Participants) | 4 | 3 | 9 | 3
  PCWP: 2 hours | -1.50 (5.000) | -3.33 (1.528) | 1.56 (3.609) | -0.67 (7.506)
  PCWP: 3 hours: number analyzed (Participants) | 4 | 3 | 9 | 3
  PCWP: 3 hours | -3.75 (3.594) | -0.33 (4.509) | -3.67 (3.464) | -3.67 (7.506)
  PCWP: 4 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PCWP: 4 hours | -2.75 (3.948) | -0.67 (5.033) | -2.90 (5.384) | -5.00 (9.165)
  PCWP: 5 hours: number analyzed (Participants) | 4 | 3 | 9 | 3
  PCWP: 5 hours | -0.50 (6.137) | -1.33 (6.110) | -1.56 (2.698) | -3.33 (9.018)
  PCWP: 6 hours: number analyzed (Participants) | 4 | 3 | 8 | 3
  PCWP: 6 hours | -0.75 (7.411) | -1.67 (5.686) | -1.25 (2.315) | -1.67 (9.504)
  RAP: 0.5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  RAP: 0.5 hours | 0.50 (1.291) | 0.00 (1.732) | 1.40 (3.836) | -1.33 (2.517)
  RAP: 1 hour: number analyzed (Participants) | 4 | 3 | 10 | 3
  RAP: 1 hour | 2.50 (3.317) | 0.33 (2.309) | 0.00 (2.867) | 3.33 (6.658)
  RAP: 2 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  RAP: 2 hours | 1.00 (0.816) | -1.00 (1.000) | 1.00 (4.397) | 2.67 (7.234)
  RAP: 3 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  RAP: 3 hours | -0.25 (1.258) | 0.33 (2.517) | 0.40 (2.366) | 3.33 (8.505)
  RAP: 4 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  RAP: 4 hours | -0.75 (4.500) | -0.67 (1.155) | -0.20 (4.315) | 4.00 (6.083)
  RAP: 5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  RAP: 5 hours | -1.50 (3.416) | -2.67 (1.155) | 0.50 (4.301) | 1.67 (8.327)
  RAP: 6 hours: number analyzed (Participants) | 3 | 3 | 10 | 3
  RAP: 6 hours | -0.67 (4.041) | -1.67 (1.528) | -0.50 (5.233) | 4.00 (8.660)
  PAS: 0.5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAS: 0.5 hours | 1.50 (5.196) | -1.00 (2.646) | 0.20 (6.033) | -0.67 (6.110)
  PAS: 1 hour: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAS: 1 hour | 4.50 (9.147) | -0.67 (4.041) | -1.50 (4.859) | -0.67 (6.028)
  PAS: 2 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAS: 2 hours | 6.25 (4.717) | 0.67 (0.577) | 0.90 (6.740) | 0.33 (4.933)
  PAS: 3 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAS: 3 hours | 7.25 (6.185) | 1.67 (5.033) | -1.40 (9.383) | -3.33 (9.292)
  PAS: 4 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAS: 4 hours | 5.75 (13.525) | 2.00 (4.359) | -1.70 (6.201) | -8.33 (15.631)
  PAS: 5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAS: 5 hours | 6.00 (11.195) | 5.00 (1.000) | -1.30 (6.945) | -1.33 (6.658)
  PAS: 6 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAS: 6 hours | 4.25 (9.179) | 2.67 (2.309) | -0.90 (8.569) | -4.33 (9.609)
  PAD: 0.5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAD: 0.5 hours | -1.25 (3.500) | 0.00 (0.000) | -1.00 (2.789) | 0.33 (4.509)
  PAD: 1 hour: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAD: 1 hour | 0.50 (2.646) | -1.33 (0.577) | -0.90 (3.872) | -1.67 (4.041)
  PAD: 2 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAD: 2 hours | -0.25 (2.217) | -0.67 (2.517) | -0.70 (3.860) | -1.00 (3.000)
  PAD: 3 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAD: 3 hours | -1.25 (4.193) | 1.00 (2.646) | -3.60 (5.168) | 0.00 (6.245)
  PAD: 4 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAD: 4 hours | -3.50 (8.888) | 1.33 (1.155) | -2.40 (4.061) | -3.00 (7.937)
  PAD: 5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAD: 5 hours | -2.50 (4.041) | 1.00 (2.646) | -2.40 (3.688) | 1.33 (5.033)
  PAD: 6 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAD: 6 hours | -4.00 (5.831) | 1.33 (3.215) | -1.80 (4.984) | 0.67 (5.686)

11. Secondary Outcome: Part A: Change in Pulmonary Artery Pulsatility Index (PAPi) Measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 Hours
Description: PAPi is a hemodynamic parameter that is derived from right atrial and pulmonary artery pulse pressures. PAPi = (PAS - PAD)/right atrial pressure. Change in PAPi measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 hours during the 6-hour IV infusion was reported in this outcome measure.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Ratio
  PAPi: 0.5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAPi: 0.5 hours | 0.28 (0.411) | -0.17 (0.833) | -0.11 (0.713) | 0.37 (1.343)
  PAPi: 1 hour: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAPi: 1 hour | -0.08 (0.562) | 0.17 (0.306) | -0.21 (0.835) | -0.17 (0.603)
  PAPi: 2 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAPi: 2 hours | 0.38 (0.435) | 0.33 (0.058) | -0.14 (1.011) | 0.20 (0.900)
  PAPi: 3 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAPi: 3 hours | 0.65 (0.624) | 0.43 (0.777) | 0.03 (0.897) | -0.33 (0.611)
  PAPi: 4 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAPi: 4 hours | 1.35 (1.838) | 0.83 (1.834) | 0.27 (1.203) | -1.03 (0.907)
  PAPi: 5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  PAPi: 5 hours | 0.95 (0.597) | 2.33 (1.818) | -0.01 (0.872) | 0.87 (2.639)
  PAPi: 6 hours: number analyzed (Participants) | 3 | 3 | 10 | 3
  PAPi: 6 hours | 0.93 (0.929) | 1.27 (0.929) | 0.77 (2.470) | -0.90 (0.173)

12. Secondary Outcome: Part A: Change in Systemic Vascular Resistance Measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 Hours
Description: Systemic vascular resistance (SVR) is the amount of force exerted on circulating blood by the vasculature of the body. SVR was calculated as 80*(mean arterial pressure - mean venous pressure) divided by cardiac output. Change in SVR measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 hours during the 6-hour IV infusion was reported in this outcome measure.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Millimeter of mercury*minutes/milliliter
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Millimeter of mercury*minutes/milliliter
  SVR: 0.5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVR: 0.5 hours | 10.30 (74.776) | -71.27 (55.492) | -47.30 (139.874) | 74.13 (198.427)
  SVR: 1 hour: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVR: 1 hour | -80.50 (57.295) | -86.30 (80.694) | 16.71 (231.657) | -131.93 (91.886)
  SVR: 2 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVR: 2 hours | -48.83 (71.811) | -46.23 (28.762) | -42.16 (205.772) | -49.40 (136.124)
  SVR: 3 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVR: 3 hours | -67.63 (56.169) | -8.10 (102.327) | -101.20 (188.863) | -195.77 (101.041)
  SVR: 4 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVR: 4 hours | -27.20 (104.351) | 73.90 (136.245) | -33.91 (241.040) | -311.03 (145.094)
  SVR: 5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVR: 5 hours | 21.10 (112.824) | 132.63 (171.630) | -92.29 (94.834) | -110.57 (222.498)
  SVR: 6 hours: number analyzed (Participants) | 3 | 3 | 10 | 3
  SVR: 6 hours | 33.10 (106.652) | 90.37 (137.576) | -70.00 (116.681) | -104.23 (90.537)

13. Secondary Outcome: Part A: Change in Systemic Vascular Resistance Index (SVRI) Measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 Hours
Description: SVRI was calculated by dividing the difference between mean arterial pressure and central venous pressure by cardiac index and multiplying by 80. Change in SVRI measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 hours during the 6 hour IV infusion was reported in this outcome measure.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Dynes*second*meter^2 per centimeter^5
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Dynes*second*meter^2 per centimeter^5
  SVRI: 0.5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVRI: 0.5 hours | 5.00 (157.514) | -171.20 (154.962) | -98.41 (270.327) | 107.83 (428.022)
  SVRI: 1 hour: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVRI: 1 hour | -156.58 (105.011) | -202.73 (185.527) | 16.20 (404.144) | -289.57 (102.838)
  SVRI: 2 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVRI: 2 hours | -115.13 (165.795) | -85.30 (63.286) | -94.82 (407.893) | -64.77 (281.682)
  SVRI: 3 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVRI: 3 hours | -152.98 (108.934) | -42.57 (192.932) | -190.53 (315.500) | -403.47 (271.919)
  SVRI: 4 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVRI: 4 hours | -85.05 (224.198) | 201.20 (357.587) | -31.66 (414.786) | -649.80 (360.988)
  SVRI: 5 hours: number analyzed (Participants) | 4 | 3 | 10 | 3
  SVRI: 5 hours | 12.80 (208.554) | 350.47 (458.646) | -172.77 (186.678) | -260.83 (484.601)
  SVRI: 6 hours: number analyzed (Participants) | 3 | 3 | 10 | 3
  SVRI: 6 hours | 61.47 (205.227) | 152.63 (171.695) | -94.08 (306.599) | -227.17 (126.337)

14. Secondary Outcome: Part A: Change in Pulmonary Vascular Resistance (PVR) Measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 Hours
Description: PVR is the resistance against blood flow from the pulmonary artery to the left atrium. Change in PVR measured by RHC at 0.5, 1, 2, 3, 4, 5 and 6 hours during the 6 hour IV infusion was reported in this outcome measure.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: dynes*second per centimeter^5
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
dynes*second per centimeter^5
  PVR: 0.5 hours: number analyzed (Participants) | 4 | 3 | 9 | 3
  PVR: 0.5 hours | -28.98 (21.955) | -97.13 (134.474) | 14.83 (115.974) | 83.40 (80.442)
  PVR: 1 hour: number analyzed (Participants) | 4 | 3 | 9 | 3
  PVR: 1 hour | 5.80 (108.571) | -37.57 (102.284) | 78.37 (235.884) | 6.40 (115.783)
  PVR: 2 hours: number analyzed (Participants) | 4 | 3 | 9 | 3
  PVR: 2 hours | 37.68 (106.364) | 46.43 (27.918) | -1.64 (290.121) | -0.10 (136.989)
  PVR: 3 hours: number analyzed (Participants) | 4 | 3 | 9 | 3
  PVR: 3 hours | 29.70 (99.607) | -11.60 (69.295) | 36.04 (171.091) | 18.13 (107.316)
  PVR: 4 hours: number analyzed (Participants) | 4 | 3 | 9 | 3
  PVR: 4 hours | 32.28 (190.279) | 10.03 (72.673) | 32.44 (191.341) | -44.03 (121.310)
  PVR: 5 hours: number analyzed (Participants) | 4 | 3 | 9 | 3
  PVR: 5 hours | 29.08 (163.825) | 44.57 (38.099) | 22.61 (195.626) | 53.70 (211.590)
  PVR: 6 hours: number analyzed (Participants) | 4 | 3 | 8 | 3
  PVR: 6 hours | 2.70 (150.529) | 54.57 (15.245) | 38.10 (291.188) | 19.53 (86.649)

15. Secondary Outcome: Part A: Change in Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and Mean Arterial Pressure (MAP) at 0.5, 1, 2, 3, 4, 5 and 6 Hours
Description: SBP, DBP and MAP were measured in a supine or seated position after participant had at least 5 minutes of rest. MAP is the average pressure of the blood circulating through a participant's arteries during the cardiac cycle. MAP was derived by using the following formula: DBP + 1/3(SBP-DBP).
Time Frame: as for outcome 9
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Millimeters of mercury
  SBP: 0.5 hours | 7.3 (10.21) | -11.0 (10.15) | -2.2 (11.47) | -0.5 (6.35)
  SBP: 1 hour | 6.8 (10.56) | -7.3 (1.53) | -3.8 (9.44) | -0.8 (6.18)
  SBP: 2 hours | 8.0 (14.54) | -6.3 (9.81) | -2.6 (11.21) | 0.5 (6.14)
  SBP: 3 hours | -1.0 (14.07) | -4.7 (7.77) | -3.9 (10.35) | -1.0 (10.30)
  SBP: 4 hours | 2.5 (15.11) | -2.7 (8.33) | -3.9 (9.66) | 0.5 (14.93)
  SBP: 6 hours | 9.8 (12.45) | -5.0 (6.00) | -1.4 (8.90) | -1.0 (12.57)
  DBP: 0.5 hours | 3.0 (16.06) | -6.7 (7.02) | -0.2 (4.92) | 0.0 (4.24)
  DBP: 1 hour | 3.0 (14.85) | -4.0 (5.29) | -2.2 (5.74) | 7.0 (18.20)
  DBP: 2 hours | 10.0 (16.12) | -7.0 (2.65) | 0.0 (7.92) | -1.5 (5.92)
  DBP: 3 hours | -4.0 (12.46) | -3.3 (5.13) | -4.8 (9.26) | -1.0 (7.79)
  DBP: 4 hours | -2.8 (13.10) | 0.3 (7.77) | -6.3 (5.76) | -1.0 (5.72)
  DBP: 5 hours | -0.8 (13.67) | -2.0 (1.73) | -6.8 (6.52) | -1.0 (6.98)
  DBP: 6 hours | 1.3 (13.57) | 1.3 (2.08) | -0.3 (6.87) | 3.8 (7.93)
  MAP: 0.5 hours | 4.42 (13.723) | -8.11 (8.002) | -0.85 (4.994) | -0.17 (4.041)
  MAP: 1 hour | 4.25 (12.971) | -5.11 (3.097) | -2.73 (4.718) | 4.42 (10.651)
  MAP: 2 hours | 9.33 (13.891) | -6.78 (4.623) | -0.88 (6.634) | -0.83 (5.828)
  MAP: 3 hours | -3.00 (12.640) | -3.78 (5.274) | -4.52 (7.752) | -1.00 (8.551)
  MAP: 4 hours | -1.00 (13.101) | -0.67 (6.960) | -5.48 (5.768) | -0.50 (8.131)
  MAP: 5 hours | 1.33 (13.570) | -1.00 (5.196) | -7.30 (5.742) | -0.17 (7.466)
  MAP: 6 hours | 4.08 (12.900) | -0.78 (1.388) | -0.64 (5.934) | 2.17 (9.406)

16. Secondary Outcome: Part A: Change in Heart Rate at 0.5, 1, 2, 3, 4, 5 and 6 Hours
Description: Heart rate was measured in a supine or seated position after participant had at least 5 minutes of rest.
Time Frame: as for outcome 9
Population: Full analysis set included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Beats per minute
  0.5 hours | -8.8 (9.00) | -7.3 (12.66) | 0.0 (5.93) | 3.5 (9.11)
  1 hour | -2.5 (2.65) | -3.3 (14.19) | -1.6 (4.86) | -9.0 (13.29)
  2 hours | -2.3 (5.32) | -0.7 (9.07) | -1.5 (6.62) | -7.0 (13.49)
  3 hours | 2.0 (8.87) | 0.0 (9.17) | -0.6 (8.31) | -5.3 (11.18)
  4 hours | -0.5 (6.24) | 0.3 (14.22) | -1.1 (5.80) | 1.0 (20.02)
  5 hours | -6.3 (6.08) | -1.7 (5.86) | -1.5 (5.77) | -5.0 (13.49)
  6 hours | 4.5 (9.00) | 1.0 (5.57) | 4.2 (9.22) | -1.5 (17.82)

17. Secondary Outcome: Part A: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence that did not necessarily have a causal relationship with study treatment. TEAEs were defined as those AEs with onset after start date/timepoint of study drug administration.
Time Frame: From start of study treatment on Day 1 up to Day 9
Population: Safety set included all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
Number analyzed (Participants) | 4 | 3 | 11 | 4
Participants | 1 | 1 | 3 | 1

18. Secondary Outcome: Part A: Area Under the Plasma Concentration Time Curve From Time Zero to 6 Hours (AUC[0-6]) of APD418
Description: AUC [0-6] was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6 hours post infusion start
Population: Pharmacokinetic (PK) set included all participants in the safety set with at least 1 post-dose PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 11
Hours*nanogram per milliliter | 6620 (68.7) | 5970 (268)

19. Secondary Outcome: Part A: Area Under the Plasma Concentration Time Curve From Time Zero to Last Quantifiable Plasma Concentration (AUCLast) of APD418
Description: AUClast was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 6.083, 6.167, 6.25, 6.5, 7, 8, 10, 18 and 24 hours post infusion start
Population: PK set included all participants in the safety set with at least 1 post-dose PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 11
Hours*nanogram per milliliter | 9410 (84.3) | 9230 (164)

20. Secondary Outcome: Part A: Area Under the Plasma Concentration Time Curve From Time Zero up to Infinity (AUC[0-Infinity]) of APD418
Description: AUC [0-infinity] was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 6.083, 6.167, 6.25, 6.5, 7, 8, 10, 18 and 24 hours post infusion start
Population: PK set included all participants in the safety set with at least 1 post-dose PK measurement. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 9
Hours*nanogram per milliliter | 9660 (87.0) | 13400 (34.5)

21. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of APD418
Description: Cmax of APD418 was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 6.083, 6.167, 6.25, 6.5, 7, 8, 10, 18 and 24 hours post infusion start
Population: PK set included all participants in the safety set with at least 1 post-dose PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 11
Nanogram per milliliter | 1540 (88.8) | 1480 (277)

22. Secondary Outcome: Part A: Terminal Elimination Half-Life (t1/2) for APD418
Description: Terminal t1/2 of APD418 was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 6.083, 6.167, 6.25, 6.5, 7, 8, 10, 18 and 24 hours post infusion start
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 9
Hours | 5.26 (0.960) | 5.26 (0.998)

23. Secondary Outcome: Part A: Distributional Half-Life (t1/2a) for APD418
Description: Distributional t1/2 of APD418 was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 6.083, 6.167, 6.25, 6.5, 7, 8, 10, 18 and 24 hours post infusion start
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 3 | 9
Hours | 0.579 (0.381) | 0.381 (0.119)

24. Secondary Outcome: Part A: Time to Maximum Observed Plasma Concentration (Tmax) for APD418
Description: Tmax of APD418 was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 6.083, 6.167, 6.25, 6.5, 7, 8, 10, 18 and 24 hours post infusion start
Population: PK set included all participants in the safety set with at least 1 post-dose PK measurement.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 11
Hours | 5.42 [4.00 to 6.08] | 5.00 [0.500 to 6.18]

25. Secondary Outcome: Part A: Total Clearance (CL) for APD418
Description: IV CL of APD418 was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 6.083, 6.167, 6.25, 6.5, 7, 8, 10, 18 and 24 hours post infusion start
Population: The PK set included all participants in the safety set with at least 1 post-dose PK measurement. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 9
Liter per hour | 9.16 (92.7) | 17.8 (23.2)

26. Secondary Outcome: Part A: Total Volume of Distribution Based on the Terminal Phase (Vdz) for APD418
Description: Vdz of APD418 was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 6.083, 6.167, 6.25, 6.5, 7, 8, 10, 18 and 24 hours post infusion start
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 9
Liter | 68.6 (74.5) | 133 (28.6)

27. Secondary Outcome: Part A: Volume of Distribution at Steady State (Vdss) for APD418
Description: Vdss of APD418 was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 6.083, 6.167, 6.25, 6.5, 7, 8, 10, 18 and 24 hours post infusion start
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 9
Liter | 27.7 (42.2) | 46.0 (34.5)

28. Secondary Outcome: Part A: Mean Residence Time From Time Zero to Time of Last Quantifiable Plasma Concentration (MRTlast) for APD418
Description: MRTlast of APD418 was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 6.083, 6.167, 6.25, 6.5, 7, 8, 10, 18 and 24 hours post infusion start
Population: PK set included all participants in the safety set with at least 1 post-dose PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 11
Hours | 2.44 (33.6) | 2.54 (74.3)

29. Secondary Outcome: Part A: Average Plasma Concentration During Dosing Interval (Cave) for ADP418
Description: Average plasma concentration calculated over the 6-hour infusion time was reported in this outcome measure.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6 hours post infusion start
Population: PK set included all participants in the safety set with at least 1 post-dose PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 11
Nanogram per milliliter | 1100 (68.7) | 996 (268)

30. Secondary Outcome: Part A: Renal Clearance (CLr) for ADP418
Description: CLr for APD418 was reported in this outcome measure.
Time Frame: Pre-dose (0) to 24 hours post infusion start, collected over 0 to 6 hour, 6 to 10 hour and 10 to 24-hour intervals
Population: PK set included all participants in the safety set with at least 1 post-dose PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 11
Liter per hour | 2.14 (55.3) | 3.78 (54.8)

31. Other Pre Specified Outcome: Part A: Amount of Unchanged Drug Excreted in Urine During Each Collection Interval From t1 to t2 (Aet1-t2)
Description: Amount of unchanged drug excreted in urine during each collection interval from t1 to t2 was reported in this outcome measure.
Time Frame: Anytime between 0 to 6 hours, 6 to 10 hours and 10 to 24 hours post infusion start
Population: PK set included all participants in the safety set with at least 1 post-dose PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 11
Milligrams
  Ae 0-6 | 11.8 (26.7) | 25.6 (56.9)
  Ae 6-10 | 4.47 (27.3) | 7.68 (68.4)
  Ae 10-24 | 2.83 (136) | 7.93 (172)

32. Other Pre Specified Outcome: Part A: Total Amount of Unchanged Drug Excreted in Urine Over the Collection Period (Amount Excreted [Ae])
Description: Total amount of unchanged drug excreted in urine over the collection period was reported in this outcome measure.
Time Frame: Pre-dose (0) to 24 hours post infusion start, collected over 0 to 6 hour, 6 to 10 hour and 10 to 24-hour intervals
Population: PK set included all participants in the safety set with at least 1 post-dose PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 11
Milligrams | 20.1 (28.8) | 48.5 (38.0)

33. Other Pre Specified Outcome: Part A: Fraction of Drug Excreted Unchanged (Fe) in Urine
Description: Fraction of drug excreted in urine was reported in this outcome measure. Data is presented in terms of percentages.
Time Frame: Pre-dose (0) to 24 hours post infusion start, collected over 0 to 6 hour, 6 to 10 hour and 10 to 24-hour intervals
Population: PK set included all participants in the safety set with at least 1 post-dose PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of unchanged drug
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 2- 0.5 mg/kg/hr APD418
Number analyzed (Participants) | 4 | 11
Percentage of unchanged drug | 22.7 (31.2) | 19.7 (39.8)

ADVERSE EVENTS:
Time Frame: From start of study treatment on Day 1 up to Day 9
Description: Safety set included all randomized participants who received at least one dose of study treatment.
Arm/Group | Cohort 1- 0.17 mg/kg/hr APD418 | Cohort 1- Placebo | Cohort 2- 0.5 mg/kg/hr APD418 | Cohort 2- Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/11 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/11 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 1/3 | 3/11 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1- 0.17 mg/kg/hr APD418 (N=4) | Cohort 1- Placebo (N=3) | Cohort 2- 0.5 mg/kg/hr APD418 (N=11) | Cohort 2- Placebo (N=4)
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Vein rupture (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early due to a business decision that was not due to any safety concerns. The number of participants was smaller than originally planned and only summary statistics were therefore generated for primary and secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT05139615/Prot_SAP_000.pdf